CLINICAL TRIAL: NCT06233760
Title: Prevalence of Abuse Among Patients With Rheumatic Diseases
Status: Recruiting | Type: Observational
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Virginia Pascual Ramos, Principal investigator, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Other Study IDs: IRE3234
Record Dates: First submitted 2024-01-14; First posted 2024-01-31 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Rheumatic Diseases; Abuse Neglect; Abuse
Keywords: rheumatic diseases; Abuse
MeSH Terms: conditions — Rheumatic Diseases | interventions — ametantrone

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with rheumatic diseases: All the rheumatic diseases outpatients from the National Institute of Medical Sciences
  Interventions: Other: Rheumatic diseases Mistreatment Scale (RDMS); Other: Health Assessment Questionnaire (HAQ); Other: Depression, Anxiety and Stress Scale (DASS-21); Other: Brief Resilient Coping Scale; Other: WHOQOL-BREF; Other: Routine assessment of patient index data 3 (RAPID-3); Other: Big Five Inventory; Other: Family APGAR Questionnaire

INTERVENTIONS:
Other: Rheumatic diseases Mistreatment Scale (RDMS) — In 2012 Giraldo-Rodríguez developed and validated the Geriatric Mistreatment Scale (GAS), prior to its application, translation, cultural adaptation, and validation were performed.
  Other Names: RD-MS
Other: Health Assessment Questionnaire (HAQ) — The HAQ is based on five patient-centered dimensions: disability, pain, medication effects, costs of care, and mortality
  Other Names: HAQ
Other: Depression, Anxiety and Stress Scale (DASS-21) — DASS-21 is a set of three self-report scales designed to measure the emotional states of depression, anxiety, and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content
  Other Names: DASS-21
Other: Brief Resilient Coping Scale — Brief Resilient Coping Scale is a 4-item measure designed to capture tendencies to cope with stress in a highly adaptive manner
  Other Names: BRCS
Other: WHOQOL-BREF — WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health, psychological health, social relationships, and environmental health; it also contains QOL and general health items
Other: Routine assessment of patient index data 3 (RAPID-3) — RAPID- 3 measures: function, pain, and patient global estimate of status. Each of the 3 individual measures is scored 0 to 10, for a total of 30
  Other Names: RAPID-3
Other: Big Five Inventory — The BFI-10 is a 10-item scale measuring the Big Five personality traits Extraversion, Agreeableness, Conscientiousness, Emotional Stability, and Openness.
  Other Names: BFI-10
Other: Family APGAR Questionnaire — Family APGAR questionnaire is used to evaluate family function, in the context of family medical care
  Other Names: APGAR

SUMMARY:
Patients with rheumatic diseases (RD) have a relevant representation in the adult population in Mexico. RD are characterized by their chronic and progressive nature, which can impact functionality during the disease and can present various factors that can be associated with the presence of abuse, among others, economic dependence, decreased physical capacity, and need for care and support in different health processes.

Regarding abuse in patients with RD, there is little information in the literature; however, it is possible that the prevalence could be similar to that of the occurrence in older adults since both populations share important states of vulnerability.

The study aimed to identify the prevalence of abuse in patients with RD. The study will be conducted in two phases: the first one in which the GAS will be adapted for patients with RD, and this version will be validated in a population of our Institute, and the second one in which, applying the validated instrument, the magnitude of abuse is evaluated, and the factors associated with this phenomenon among patients with RD are explored.

DETAILED DESCRIPTION:
Patients with rheumatic diseases (RD) have a relevant representation in the adult population in Mexico. RD are characterized by their chronic and progressive nature, which can impact functionality during the disease and can present various factors that can be associated with the presence of abuse, among others, economic dependence, decreased physical capacity, and need for care and support in different health processes.

In 1970, the phenomenon of abuse in geriatric patients was described for the first time as a phenomenon identified as a public health problem and an issue of human rights violation.

In 2012 Giraldo-Rodríguez developed and validated the Geriatric Abuse Scale (GAS), an instrument that, with adequate psychometric properties, reported a prevalence of abuse of 10.28% in Mexico.

Regarding abuse in patients with RD, there is little information in the literature; however, it is possible that the prevalence could be similar to that of the occurrence in older adults since both populations share important states of vulnerability.

The study aimed to identify the prevalence of abuse in patients with RD. The study will be conducted in two phases: the first one in which the GAS will be adapted for patients with RD, and this version will be validated in a population of our Institute, and the second one in which, applying the validated instrument, the magnitude of abuse is evaluated, and the factors associated with this phenomenon among patients with RD are explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a rheumatic disease diagnosis according to their primary rheumatologist who agree to participate

Exclusion Criteria:

* Patients with a not confirmed rheumatic disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the rheumatic diseases outpatients from the National Institute of Medical Sciences
Sampling Method: Probability Sample
Enrollment: 244 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Number of Mexican patients with RD who will present the phenomenon of mistreatment | At inclusion (baseline moment) (cross-sectional study)
  Identify the percentage of patients with rheumatic diseases that present mistreatment using the instrument developed by Giraldo-Rodríguez et al (translation, cultural adaptation, and validation performed)

SECONDARY OUTCOMES:
Identify factors associated with mistreatment among patients with rheumatic diseases | At inclusion (baseline moment) (cross-sectional study)
  Identify factors associated with mistreatment among patients with rheumatic diseases using an instrument locally development

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Dr Pascual-Ramos, Principal Investigator — INNSZ
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giraldo-Rodriguez L, Rosas-Carrasco O. Development and psychometric properties of the Geriatric Mistreatment Scale. Geriatr Gerontol Int. 2013 Apr;13(2):466-74. doi: 10.1111/j.1447-0594.2012.00894.x. Epub 2012 Jun 14. PMID 22694594
- [Background] Castro I, Barrantes F, Tuna M, Cabrera G, Garcia C, Recinos M, Espinoza LR, Garcia-Kutzbach A. Prevalence of abuse in fibromyalgia and other rheumatic disorders at a specialized clinic in rheumatic diseases in Guatemala City. J Clin Rheumatol. 2005 Jun;11(3):140-5. doi: 10.1097/01.rhu.0000164823.78761.a2. PMID 16357732